CLINICAL TRIAL: NCT04638283
Title: The Efficacy of Goal Focused, Non-Pharmacological Treatment for Persons With ADHD/ADD. A Randomized Controlled Trial.
Brief Title: The Efficacy of Goal Focused, Non-Pharmacological Treatment for Persons With ADHD/ADD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Kjersti Traeland Hanssen, PhD/Clinical neuropsychologist, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Goal Focused ADHD Treatment
Record Dates: First submitted 2020-10-15; First posted 2020-11-20 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Attention-Deficit Hyperactivity Disorder, Unspecified Type
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The participant is randomized by a lottery to participate either in the intervention group receiving the intervention described above or the controlgroup receiving TAU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventioh group (Experimental): The intervention consists of
  1. Eight group sessions of two hours duration, focusing on GMT and ADHD. The Group consists of six participants and is directed by one neuropsychologist and one psychologist.
  2. Four individual sessions with the neuropsychologist/psychologist directing the Group where the participant is guided through the process of formulating GAS-goals.
  3. Bi-weekly Telephone follow up focusing on GAS-goal attainment the thre first months following the Group session phase.
  Interventions: Behavioral: Goal Attainment Scaling
- Control Group (No Intervention): Participants in the Control Group receive TAU. Participation in the study does not influence decisions regarding pharmacological interventions in either of the groups.

INTERVENTIONS:
Behavioral: Goal Attainment Scaling — Individual goals will be formulated and measured by Goal Attainment Scaling (GAS). GAS provides a method for quantifying the attainment of individualized goals, typically set in cognitive rehabilitation. Different levels of outcomes for each goal are operationalized in a five-point scale and given a numeric value. For each individual goal, minus two refers to the goal attainment much less than expected, minus one refers to a little less than expected, zero refers to expected outcome, plus one refers to a little bit better than expected and plus two refers to goal attainment much better than expected. The participants can establish as many goals as desired. Outcomes can be summed within different patient goals, as well as across patients to assess overall outcome of treatment outcomes.
  Arms: Interventioh group

SUMMARY:
The study aims to improve the understanding of non-pharmacological treatments of ADHD with a particular emphasis on coping with executive problems. Executive functions can be defined as those abilities necessary to formulate goals, carry them out effectively and enabling a person to engage successfully in independent, purposive, self-serving behavior.

The intervention consists of:

1. Eight psycho-educative group sessions focusing on Goal Management Training (GMT), a method aiming to enhance goal directed behavior, developed by Levine and colleagues in 2011.
2. Four individual sessions where the participants are guided through the process of formulation individual goals for improving functioning in everyday life. The method used for goal setting is Goal Attainment Scaling (GAS), developed by Kiresuk and Sherman in 1968.
3. Bi-weekly telephone follow up the first three months preceding the group sessions, focusing on the attainment of GAS-goals.

Adult participants with ADHD/ADD are recruited from the outpatient psychiatric health care clinic, DPS Nedre Romerike at Akershus University Hospital and are randomized into either 1) an intervention-group, receiving the intervention described above or 2) a control-group receiving treatment as usual.

It is hypothesized that the intervention will improve executive functioning, reported ADHD-symptoms and psychological well-being. It is also hypothesized that the participants sucessfully will formulate and implement GAS-goals and that goal attainment will sustain throughout the follow-up phase.

DETAILED DESCRIPTION:
Given the 1) high prevalence and possible detrimental consequences of ADHD, 2) limitations related to pharmacological ADHD-treatments, 3) scarce evidence of the effects of long term use of pharmacological treatment and 4) limitations related to the present evidence base for the effects of non-pharmacological treatments, research on the effects of non-pharmacological ADHD treatment is highly required.

Goal Management Training (GMT) (Levine et al, 2011) is a theory-driven intervention relying on metacognitive strategies to reengage endogenous attention processes, in addition to teaching problem-solving techniques to improve goal-directed capacity. GMT draws upon theories regarding sustained attention, mindfulness and goal processing. The aim is to increase awareness of errors and strategies while facing complex, everyday challenges. The patient learns to stop ongoing behavior, define goal hierarchies and to adjust and monitor goals. Generalization to everyday-life is heavily emphasized.

In previous studies, GMT has been shown to improve goal directed behaviour including generalization effects to daily life and psychological well-being in various neurological conditions, e.g. acquired brain injury and spina bifida (Hypher et al, 2019; Stubberud et al, 2014; Tornås et al, 2016) and normal ageing (Levine et al, 2007). The evidence of GMT in the adult ADHD populations is scarce.

To the investigators knowledge, this is the first trial combining group based, GMT and individual goal setting within the frame of a psycho-educative, cognitive rehabilitation intervention in order to help adults with ADHD cope with executive problems in everyday life.

Research questions and hypotheses

1. Does the intervention combining GMT, psychoeducation and implementation of GAS goals result in improvements in executive problems for adults with ADHD when compared to treatment as usual (TAU)? Hypothesis 1: Post intervention changes in executive functions will be reflected in improved scores on a measure pertaining to daily life executive function (BRIEF-A) at five- and eights months follow up.
2. Does the intervention result in improvements of reported ADHD symptoms when compared to TAU? Hypothesis 2: Post intervention changes in ADHD-symptoms will be reflected in improved scores on a measure pertaining to ADHD-symptoms (ASRS-v1.1) at five and eight months follow-up.
3. Does participation in the intervention improve psychological well-being when compared to TAU? Hypothesis 3: Post intervention changes in psychological well-being will be reflected in improved scores on a measure pertaining to psychological well-being (HSCL-25) at five and eight months follow-up.
4. Will the participants succeed in attaining individual GAS goals for coping with executive problems? Hypothesis 4: The participants will successfully formulate and implement GAS-goals for coping with executive problems in everyday life. Goal attainment will sustain throughout the three-month long implementation phase and sustain until the eight month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Hyperkinetic disorder, ADHD or ADD. Both patients recently diagnosed at DPS and patients previously diagnosed can be included.
2. Subjective complaints about executive problems affecting everyday life, operationalized as a score of 60 or above on BRIEF-A or as reported in the inclusion interview.
3. Motivation for working with the executive problems in order to increase coping in everyday life.
4. Adequate language skills to participate in group discussions without any need for an interpreter.

Exclusion Criteria:

1. CNS injury or disease other than hyperkinetic disorder, ADHD or ADD.
2. Ongoing substance-abuse.
3. Psychopathology that would negatively interfere with participation in the intervention, e.g. ongoing psychosis, present suicidal risk to severe to be treated in an out-patient setting or personality disorders considered to severe to be treated in a group-based out-patient setting.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function for Adults (BRIEF-A) | Change from baseline BRIEF-A at 8 months.
  BRIEF-A is a standardized informant- and self report Inventory measuring different aspects of executive functions (Rabin et al, 2006). Data (BRIEF-A self report form) is collected at baseline (T1), at 2 months (T2), at 5 months (T3) and finally at 8 months (T4). BRIEF-A informant report form is collected at baseline (T1) and at 8 months (T4).
Goal Attainment Scaling (GAS). | Change from baseline GAS at 5 months.
  Individual goal attainment will be measured by GAS (Kiresuk and Sherman, 1968). Se description in the intervention-section. GAS-goals are formulated during the individual sessions and scored during biweekly telephone calls the three first months following the last group session.

SECONDARY OUTCOMES:
Hopkins Symptom Checklist-25 (HSCL-25) | Change from baseline HSCL-25 at 8 months.
  Psychological well-being will be measured by Hopkins Symptom Checklist-25 (Derogatis, 1947). HSCL-25 is a screening instrument measuring the presence and intensity of symptoms of anxiety and depression.Data collected at baseline (T1), at 2 months (T2), at 5 months (T3) and finally at 8 months.
The Adult ADHD Self Report Scale (ASRS-v.1.1) | Change from baseline ASRS-v.1.1 at 8 months.
  ASRS-v1.1 (Kessler et al, 2005) us a questionnaire addressing symptoms of ADHD, developed in conjunction with the World Health Organization (Kessler et al, 2005). Data collected at baseline (T1), at 2 months (T2), at 5 months (T3) and finally at 8 months (T4)

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti T Hanssen, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, DPS Nedre Romerike, Postboks 1000, Loerenskog, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Adler L, Ames M, Demler O, Faraone S, Hiripi E, Howes MJ, Jin R, Secnik K, Spencer T, Ustun TB, Walters EE. The World Health Organization Adult ADHD Self-Report Scale (ASRS): a short screening scale for use in the general population. Psychol Med. 2005 Feb;35(2):245-56. doi: 10.1017/s0033291704002892. PMID 15841682
- [Background] Kiresuk TJ, Sherman RE. Goal attainment scaling: A general method for evaluating comprehensive community mental health programs. Community Ment Health J. 1968 Dec;4(6):443-53. doi: 10.1007/BF01530764. PMID 24185570
- [Background] Levine B, Schweizer TA, O'Connor C, Turner G, Gillingham S, Stuss DT, Manly T, Robertson IH. Rehabilitation of executive functioning in patients with frontal lobe brain damage with goal management training. Front Hum Neurosci. 2011 Feb 17;5:9. doi: 10.3389/fnhum.2011.00009. eCollection 2011. PMID 21369362
- [Background] Levine B, Stuss DT, Winocur G, Binns MA, Fahy L, Mandic M, Bridges K, Robertson IH. Cognitive rehabilitation in the elderly: effects on strategic behavior in relation to goal management. J Int Neuropsychol Soc. 2007 Jan;13(1):143-52. doi: 10.1017/S1355617707070178. PMID 17166313
- [Background] Rabin LA, Roth RM, Isquith PK, Wishart HA, Nutter-Upham KE, Pare N, Flashman LA, Saykin AJ. Self- and informant reports of executive function on the BRIEF-A in MCI and older adults with cognitive complaints. Arch Clin Neuropsychol. 2006 Oct;21(7):721-32. doi: 10.1016/j.acn.2006.08.004. Epub 2006 Sep 18. PMID 16979868
- [Background] Hypher RE, Brandt AE, Risnes K, Ro TB, Skovlund E, Andersson S, Finnanger TG, Stubberud J. Paediatric goal management training in patients with acquired brain injury: study protocol for a randomised controlled trial. BMJ Open. 2019 Aug 1;9(8):e029273. doi: 10.1136/bmjopen-2019-029273. PMID 31375619
- [Background] Stubberud J, Langenbahn D, Levine B, Stanghelle J, Schanke AK. Emotional health and coping in spina bifida after goal management training: a randomized controlled trial. Rehabil Psychol. 2015 Feb;60(1):1-16. doi: 10.1037/rep0000018. Epub 2014 Dec 15. PMID 25496433
- [Background] Tornas S, Lovstad M, Solbakk AK, Schanke AK, Stubberud J. Goal Management Training Combined With External Cuing as a Means to Improve Emotional Regulation, Psychological Functioning, and Quality of Life in Patients With Acquired Brain Injury: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Nov;97(11):1841-1852.e3. doi: 10.1016/j.apmr.2016.06.014. Epub 2016 Jul 15. PMID 27424292
- [Derived] Hanssen KT, Brevik EJ, Smastuen MC, Stubberud J. Improvement of anxiety in ADHD following goal-focused cognitive remediation: a randomized controlled trial. Front Psychol. 2023 Nov 17;14:1212502. doi: 10.3389/fpsyg.2023.1212502. eCollection 2023. PMID 38046113